CLINICAL TRIAL: NCT02642887
Title: Evaluation of Root Coverage Outcome Using a Modified Tunnel Approach Versus Tunnel Technique: A Randomized Clinical Trial
Brief Title: A Modified Tunnel Approach in Treatment of Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hala Helmi Hazzaa, Assistant Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Al-Azhar 11-2014
Record Dates: First submitted 2015-12-18; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Gingival Recession
Keywords: gingival recession; tunnel technique; Miller Class I and II
MeSH Terms: conditions — Gingival Recession | interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- The test group (Experimental): This group included 30 recession defects treated with mTA + SCTG
  Interventions: Procedure: mTA + SCTG
- The control group (No Intervention): This group included 30 recession defects treated with cTT + SCTG

INTERVENTIONS:
Procedure: mTA + SCTG — These recession defects will be covered by modified tunnel approach; using a full thickness flap till the level of mucogingival junction then, partial thickness flap will be applied in the vestibular mucosa. SCTG will be harvested from the palate, put on the root surface then covered by the mTA and sutured.
  Other Names: Dual approach + SCTG
  Arms: The test group

SUMMARY:
Objectives: To clinically evaluate the healing of Miller Class I and II isolated gingival recessions treated with the modified tunnel approach (mTA) versus the conventional tunnel technique (cTT) in conjunction with subepithelial connective tissue graft (SCTG).

Material and Methods: In this split-mouth study, thirty healthy patients exhibiting two isolating anterior Miller Class I and II gingival recessions were treated with mTA + SCTG and cTT + SCTG. Treatment outcomes were assessed at baseline, 3-months and 6-months postoperatively. The primary outcome was root coverage esthetic scores (RES).

DETAILED DESCRIPTION:
Various techniques have been suggested for the treatment of isolated mandibular recessions e.g., envelope, coronally advanced flaps double pedicle flap or tunneling procedures combined with laterally positioned pedicle flaps in conjunction with SCTG. Despite the fact that the mentioned techniques appear to improve root coverage, the success in terms of complete root coverage has high variability and thus it is still unknown which approach may lead to the most predictable outcomes. The limited evidence from the literature points clearly to the clinical importance of developing new concepts for predictable of isolated mandibular recessions.

The MTA is a dual flap approach; that starts with full thickness flap (avoiding papilla incision) till the level of the mucogingival junction. On reaching the level of the vestibular mucosa, a partial thickness flap is applied to undermine the base of the flap. Using this dual approach carries two main advantages: avoidance of severing the gingival blood supply through the full thickness flap, in addition to minimizing the tension on the flap tissue through using the partial thickness flap at the above-mentioned site.

In this trial, the mTA has been proposed for the surgical treatment of isolated mandibular recessions due to the following advantages: 1) it avoids vertical releasing incisions. 2) it doesn't incise the papilla, which may improve the vascularization of the area plus stabilizing the soft tissue flap. 3) it is suitable to patients with thin gingival biotype.

ELIGIBILITY:
Inclusion Criteria:

* except for chronic periodontitis, our patients were systemically free
* Two mandibular Miller Class I or II recession sites
* at least 2 mm attached gingiva.
* at least 3 mm depth of recession.

Exclusion Criteria:

* Systemic diseases.
* Smokers or formal smokers
* Pregnant or lactating females
* History of antibiotic therapy at the last 6 months
* Patients who are not willing to follow the study protocol

Ages: 29 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The change in Root Coverage Esthetic Score | Baseline, 3 months and 6 months
  This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color. It is calculated by expert operator.

SECONDARY OUTCOMES:
The change in percentage of root coverage | Baseline, 3 months and 6 months
  The percentage of root coverage will be calculated at 3 months, then 6 months.
The change in depth of gingival recession | Baseline, 3 months and 6 months.
  The change in depth of gingival recession will be calculated at baseline, 3 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hala H Hazzaa, Professor, Principal Investigator — Al-Azhar University, Faculty of Dental and Oral Medicine (Girls Branch)

REFERENCES:
- [Background] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000
- [Background] Cairo F, Cortellini P, Tonetti M, Nieri M, Mervelt J, Cincinelli S, Pini-Prato G. Coronally advanced flap with and without connective tissue graft for the treatment of single maxillary gingival recession with loss of inter-dental attachment. A randomized controlled clinical trial. J Clin Periodontol. 2012 Aug;39(8):760-8. doi: 10.1111/j.1600-051X.2012.01903.x. Epub 2012 May 28. PMID 22639845